CLINICAL TRIAL: NCT00018538
Title: Calcifidol Therapy in Men With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCO-09-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Prostate Cancer
Keywords: vitamin D; prostatic neoplasms; neoplasm recurrence
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

INTERVENTIONS:
Drug: calcifidiol

SUMMARY:
Prostate cancer is a common occurrence in the aging population, with one in ten men destined to develop the disease. 40% of patients with prostate cancer experience a recurrence after definitive treatment. This study addresses the as-yet unresolved problem of the optimal management of early recurrence as manifested by increase in the accepted marker for this disease, PSA. Vitamin D, an agent with cell-differentiating properties, has been shown to inhibit angiogenesis and cause differentiation of prostate cancer cells in the laboratory and to affect PSA favorably in clinical studies of patients with advanced prostate cancer. This study will assess the effects of vitamin D in patients with sub-clinical biochemical relapses of prostate cancer as indicated by rising PSA but low tumor burdens, with the potential for developing an approach to this problem that will delay or prevent progression.

ELIGIBILITY:
Patients will be males with three successive rises in PSA after achieving a nadir post-definitive therapy. The following criteria must be met: pathologically confirmed prostate cancer, completion of definitive treatment in the form of local external beam radiation or definitive surgery and three successive rises in PSA with no clinical evidence of disease.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Guy Howard, Ph.D; Gary Schwartz, Ph.D, MPH; James Schlesselman, Ph.D
Locations (1):
- VAMC Miami, FL, Miami, Florida, United States